CLINICAL TRIAL: NCT06455189
Title: Magnetic Resonance Fingerprinting Guided Extended Resection in Glioblastomas
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CASE1324
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Glioblastoma; Brain Tumor
Keywords: Radiation Therapy; Magnetic Resonance Fingerprinting; MRI
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly allocated in a one-to-one ratio to undergo either tumor resection with intraoperative MRF/MRI infiltration mapping guidance or with standard of care neurosurgical techniques. The investigators who assess eligibility of participants and schedule surgeries (neurosurgeons, residents, research nurse) will be masked to treatment group assignment by use of a sealed-envelope design. The treatment group assignments will be disclosed after surgery is scheduled and after written consent is obtained, usually on the day before the operation.
Who Masked: Outcomes Assessor
Masking Description: The neurosurgeons and participants will not be masked to the treatment group assignment, but the team members looking at outcome assessment will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Other): Routine standard of care process will be followed for neurosurgical guidance
  Interventions: Other: Control Group - Standard of care neurosurgical resection
- Group 2 (Experimental): The surgeon will have access to advanced MRI and MRF analysis research images during surgery and may use them for guidance, in addition to all routinely used surgical tools.
  Interventions: Procedure: MRF/MRI infiltration guidance for extended resection

INTERVENTIONS:
Other: Control Group - Standard of care neurosurgical resection — The control group will include only standard of care tools. - Standard of care neurosurgical resection will include the use of all standard neurosurgical instruments and techniques (eg, microscope, intraoperative ultrasound, 5-ALA fluorescence guided surgery and neuronavigation system).
  Arms: Group 1
Procedure: MRF/MRI infiltration guidance for extended resection — Magnetic resonance imaging, MRI, is a procedure that uses radio waves, a powerful magnet, and a computer to make a series of detailed pictures of areas inside the body
  Arms: Group 2

SUMMARY:
Magnetic resonance imaging, MRI, is a procedure that uses radio waves, a powerful magnet, and a computer to make a series of detailed pictures of areas inside the body. The goal of this study is to determine if MR fingerprinting, new way of acquiring MRI images, can help identify the extent of tumor spread in the brain, better than routine MRI images.

DETAILED DESCRIPTION:
Glioblastomas (GBs) are aggressive malignant brain tumors with a median survival of less than 15 months . Infiltration of cancer beyond the tumor margins causes recurrence in nearly 100% of GBs; however, this cannot be measured by current imaging techniques . Availability of reliable and reproducible infiltration prediction maps at initial diagnosis will open new treatment opportunities such as targeted surgery or escalated radiation therapy (RT).

On clinical contrast enhanced (CE) magnetic resonance imaging (MRI) scans, a typical GB demonstrates an enhancing mass with central necrosis and an extensive surrounding, peritumoral region with bright signal on T2-weighted(w) and FLAIR (Fluid attenuation inversion recovery) images. This bright, peritumoral T2/FLAIR region is known to contain vasogenic edema and tumor infiltration, as it is well known that GBs infiltrate beyond the enhancing tumor margins.

Since there is a clear link between extent of tumor resection and survival the challenge for neurosurgeons is maximizing resection of tumor, while avoiding neurological injury. Typically, the central region of the tumor can be safely resected with minimal risk. The challenge lies in maximal safe resection along the tumor margins as it infiltrates normal brain. MR Fingerprinting is a quantitative imaging (QI) scan developed at CWRU that provides rapid quantification of multiple tissue properties, such as T1 and T2 relaxation maps, with high reproducibility and excellent tissue characterization. Our preliminary analysis of retrospective data of 60 GB participants with MRF+MRI scans with targeted 5-aminolevulenic acid (5-ALA) tissue sampling demonstrates an AUC of 0.8 for MRF/MRI model for GBM infiltration prediction in peritumoral region .

ELIGIBILITY:
Stage I:

Inclusion criteria:

* Age > 18
* MR imaging findings suggestive of GB
* Maximal tumor diameter greater than 3 cm
* Ability to provide written informed consent
* Ability to undergo MRI scan
* Consideration for biopsy, subtotal or gross total resection.

Exclusion Criteria:

* Contraindications to MRI
* Contraindication to surgical treatment
* Prior treatment for glioblastoma

Stage II:

Inclusion Criteria:

* Age > 18
* MR imaging findings suggestive of GB
* Maximal tumor diameter greater than 3 cm
* Ability to provide written informed consent
* Ability to undergo MRI scan
* Lesions amenable to gross total resection
* Presence of peritumoral FLAIR signal abnormality beyond the area of enhancement.

Exclusion Criteria:

* Inability to undergo MRI imaging
* Participants undergoing only stereotactic biopsy or less than gross total resection
* Participants undergoing LITT
* Inability to consent for the study
* Previously treated/ recurrent glioma.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2029-06-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced serious adverse events(SAEs) at 48 hours post targeted biopsy sampling procedure | 48 hours post surgery
  Safety is defined as the absence of significant complications at 48 hours. SAEs are measured using BTM(Bayesian toxicity monitorin) algorithm
Number of participants who experienced serious adverse events(SAEs) at 30 days post targeted biopsy sampling procedure | 30 days post surgery
  Safety is defined as the absence of significant complications at 30 days. SAEs are measured using BTM(Bayesian toxicity monitorin) algorithm
Feasibility as assessed by the performance of MRF/MRI infiltration mapping guidance in surgical resection of new glioblastomas | Up to 72 hours post surgery
  Assessed by post surgical MRI scans

SECONDARY OUTCOMES:
Progression Free Survival(PFS) | 6 months
  PFS will be estimated using Kaplan-Meier method and the difference of PFS between two arms will be compared using log-rank test
Extent of resection | 1 week post surgery
  As assessed by post surgical MRI scans
Operator confidence | 1 week post surgery
Histopathological correlation | Approximately one week post surgery
Recurrence | Approximately 12 months post surgery
  As assessed by MRI scans

CONTACTS AND LOCATIONS:
Overall Officials: Chaitra Badve, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center; Tiffany Hodges, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, UH Department of Radiology, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No